CLINICAL TRIAL: NCT04975399
Title: A Phase 1, Multi-center, Open-label, Dose Finding Study of CC-92328 in Subjects With Relapsed and/or Refractory Multiple Myeloma
Brief Title: Study to Evaluate the Safety and Tolerability of CC-92328 in Participants With Relapsed and/or Refractory Multiple Myeloma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-92328-MM-001; 2020-005968-64 (EudraCT Number)
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; First-in-human; Phase 1; Relapsed or Refractory; CC-92328
MeSH Terms: conditions — Multiple Myeloma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of CC-92328 (Experimental): CC-92328 administered intravenously in 28-day cycles
  Interventions: Drug: CC-92328

INTERVENTIONS:
Drug: CC-92328 — CC-92328

SUMMARY:
This Phase 1, first-in-human (FIH), clinical study of CC-92328 will explore the safety, tolerability and preliminary biological and clinical activity of CC-92328 as a single-agent in the setting of relapsed and/or refractory multiple myeloma (R/R MM). The study will be conducted in two parts: monotherapy dose escalation (Part A) and monotherapy dose expansion (Part B).

ELIGIBILITY:
Inclusion Criteria:

Participants must satisfy the following criteria to be enrolled in the study:

1. must understand and voluntarily sign an informed consent form (ICF) prior to any study-related assessments/procedures being conducted.
2. willing and able to adhere to the study visit schedule and other protocol requirements.
3. Participant is ≥ 18 years of age the time of signing the ICF.
4. Participant has a history of multiple myeloma (MM) with relapsed and/or refractory disease who have failed or who are ineligible or intolerant to available therapies that may provide clinical benefit.
5. Have documented disease progression on or within 12 months from the last dose of their last myeloma therapy.
6. Participant must have measurable disease.
7. Participant has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
8. Females of childbearing potential (FCBP) must commit to true abstinence from heterosexual contact or agree to use at least one method of highly effective contraception without interruption from screening to at least 12 weeks after the last dose of CC-92328
9. Males must practice true abstinence or agree to use a condom
10. FCBP and males must avoid conceiving from signing the ICF, while participating in the study, during dose interruptions, and for at least 12 weeks after the last dose of CC-92328.

Exclusion Criteria:

The presence of any of the following will exclude a participant from enrollment:

1. Participant has symptomatic central nervous system involvement of MM.
2. Participant had a prior autologous stem cell transplant ≤ 90 days prior to starting CC-92328.
3. Participant had a prior allogeneic stem cell transplant with either standard or reduced intensity conditioning ≤ 12 months prior to starting CC-92328.
4. Participant had prior systemic cancer-directed treatments or investigational modalities ≤ 5 half-lives or 4 weeks prior to starting CC-92328, whichever is shorter.
5. Participant is a pregnant or lactating female.
6. Participant received live virus vaccines within at least 4 weeks prior to starting study drug.
7. Participant has known active human immunodeficiency virus (HIV) infection.
8. Participant has active hepatitis B or C (HBV/HCV) infection.
9. Participant weight is ≤ 40 kg at screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2024-06-18 (Actual); Study Completion 2024-06-18 (Actual)

PRIMARY OUTCOMES:
Dose-Limiting Toxicities (DLTs) | Up to 28 days after the first dose
  Are defined as toxicities that meet the protocol-specified criteria occurring within the DLT assessment window (Cycle 1, Days 1 to 28) except those that are clearly and incontrovertibly due to the underlying disease or extraneous causes.
Maximum Tolerated Dose (MTD) | Up to 12 weeks after the last dose
  Defined as the highest dose at which less than 33% of the population treated with CC-92328 experience a dose-limiting toxicity (DLT) in the first cycle and at least 6 evaluable participants have been treated at this dose level.
Incidence of Adverse Events (AEs) | Up to 12 weeks after the last dose
  Type, frequency, seriousness, severity and relationship of AEs to CC-92328.

SECONDARY OUTCOMES:
Preliminary Efficacy - Overall Response Rate (ORR) | Up to approximately 2 years
  Defined as the proportion of participants who achieve a partial response (PR) or better according to IMWG response criteria.
Preliminary Efficacy - Time to response | Up to approximately 2 years
  Defined as the time from the first CC-92328 dose date to the date of first documented response (PR or better).
Preliminary Efficacy - Duration of response | Up to approximately 2 years
  Defined as the time from the earliest date of documented response (≥ PR) to the first documented disease progression or death, whichever occurs first.
Preliminary Efficacy - Progression-free Survival (PFS) | Up to approximately 2 years
  Defined as the time from the first dose of CC-92328 to pharmacodynamics (PD) or death from any cause, whichever occurs first.
Preliminary Efficacy - Overall Survival (OS) | Up to approximately 2 years
  Defined as the time from the first dose of CC-92328 to death from any cause.
Pharmacokinetics - Cmax | Day 1 to 9 weeks after last dose of study drug
  Maximum serum concentration of drug.
Pharmacokinetics - Cmin | Day 1 to 9 weeks after last dose of study drug
  Minimum serum concentration of drug.
Pharmacokinetics - AUC | Day 1 to 9 weeks after last dose of study drug
  Area under the curve.
Pharmacokinetics - tmax | Day 1 to 9 weeks after last dose of study drug
  Time to peak (maximum) serum concentration.
Pharmacokinetics - t1/2 | Day 1 to 9 weeks after last dose of study drug
  Half-life.
Pharmacokinetics - CL | Day 1 to 9 weeks after last dose of study drug
  Total body clearance of the drug from the serum.
Pharmacokinetics - Vd | Day 1 to 9 weeks after last dose of study drug
  Volume of distribution.
Pharmacokinetics - Accumulation index of CC-92328 | Day 1 to 9 weeks after last dose of study drug
  Calculated from the serum concentration-time data of CC-92328 using non-compartment methods.
Presence of Anti-CC92328 antibodies (ADA) | Day 1 to 9 weeks after last dose of study drug
  Determined using a validated bridging immunoassay with electrochemiluminescence detection.
Frequency of Anti-CC92328 antibodies (ADA) | Day 1 to 9 weeks after last dose of study drug
  Determined using a validated bridging immunoassay with electrochemiluminescence detection.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (15):
- United States (6):
  - Local Institution - 104, Birmingham, Alabama
  - Local Institution - 105, Scottsdale, Arizona
  - Local Institution - 106, Tampa, Florida
  - Local Institution - 108, New York, New York
  - Local Institution - 107, New York, New York
  - Local Institution - 101, Milwaukee, Wisconsin
- Canada (5):
  - Local Institution - 201, Calgary, Alberta
  - Local Institution - 204, Edmonton, Alberta
  - Local Institution - 203, Halifax, Nova Scotia
  - Local Institution - 202, Toronto, Ontario
  - Local Institution - 205, Montreal, Quebec
- Spain (4):
  - Local Institution - 302, Pamplona, Navarre
  - Local Institution - 301, Badalona
  - Local Institution - 303, Salamanca
  - Local Institution - 304, Santander

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link:
  https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.celgene.com/research-development/clinical-trials/clinical-trials-data-sharing/

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSClinicalTrials.com